CLINICAL TRIAL: NCT00232453
Title: A Phase II Protocol of Preoperative Combined Radiation and Chemotherapy for Resectable Primary Rectal Cancer
Brief Title: Preoperative Combined Radiation and Chemotherapy - Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0024-C
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy

INTERVENTIONS:
Procedure: Combined Radiation and Chemotherapy

SUMMARY:
There is no established standard preoperative treatment in rectal cancer. Two large randomized studies in North America closed from lack of accrual; therefore the only method of assessing preoperative treatment in rectal cancer is from Phase II studies. This study builds on the experience at PMH gained in two previous studies which demonstrated a lower than expected toxicity with concurrent 5FU infusion and external radiotherapy. The current standard at PMH is preoperative radiation, 46Gy in 23 fractions with concurrent 5FU infusion 225mg/m2. An increase of radiation dose and consequent increase in chemotherapy may improve the response rate, but may also increase toxicity. It is proposed to increase the dose of radiotherapy to 50Gy in 25 fractions with concurrent chemotherapy and measure acute toxicity and complete remission rate.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum
* Performance status <2 (ECOG, appendix II)
* Clinical Stage T2 N1-2, T3-4 NO-2, without evidence of distant metastasis

Exclusion Criteria:

* Prior pelvic irradiation
* Inflammatory bowel disease
* Evidence of distant metastasis
* Performance status >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2001-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Assess acute toxicity and complete remission rate of combined preoperative radiation and chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: James Brierley, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network Princess Margaret Hospital, Toronto, Ontario, Canada